CLINICAL TRIAL: NCT05049265
Title: A Phase Ia Study to Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single-dose and Multiple-dose Of JS007 Injection In Patients With Advanced Solid Tumors
Brief Title: Clinical Study of JS007 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS007-001-I
Record Dates: First submitted 2021-08-19; First posted 2021-09-20 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-08

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS007 (Experimental)
  Interventions: Biological: JS007

INTERVENTIONS:
Biological: JS007 — JS007 only

SUMMARY:
This is an open label, phase Ia clinical study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, pharmacodynamic (PD) profile, immunogenicity and preliminary efficacy of JS007 in the patients with advanced solid tumors who have progressed after standard of care, or lack of effective standard therapeutic regimen. This study is divided into two periods: dose escalation period, dose expansion period.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients with age of 18~75 years;
2. Signed informed consent form;
3. Confirmed histological or cytological diagnosis of advanced or recurrent solid tumor with previous standard therapy failure, no available standard therapy or refusal of standard therapy;
4. Consent to provide tumor tissue (FFPE archival sample within 2 years, or newly obtained tissue blocks, or unstained slides from FFPE);
5. Having at least one measurable lesion in accordance with the response evaluation criteria in solid tumors (RECIST V1.1).
6. Life expectancy ≥ 3 months;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0 or 1 (Appendix 1);
8. Functional indicators of organs must fulfill the following criteria:

   i. White blood cell ≥ 2.5 × 109/L ii. Neutrophils ≥ 1.5 × 109/L iii. Platelets ≥ 85 × 109/L iv. Hemoglobin ≥ 90 g/L v. Blood creatinine ≤ 1.5 × ULN, or creatinine clearance > 40 ml/min (calculated according to Cockcroft-Gault formula, see Appendix) vi. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN (for known liver metastases: AST and ALT ≤ 5×ULN) vii. Total bilirubin ≤ 1.5 × ULN (For subjects with Gilbert's Syndrome or known liver metastases, ≤ 2×ULN is acceptable)

Exclusion criteria:

1. The patient with metastasis to the central nervous system (CNS);
2. The patient requires systemic steroids or anti-convulsant drugs, or patients with risk of intracerebral hemorrhage judged by the investigator;
3. Patients with primary CNS tumor or meningeal metastasis;
4. Having used systemic anticancer therapy, including radiotherapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy, within 4 weeks prior to the first dose, or all adverse events except hair loss have not recovered to CTCAE Grade 1 or below;
5. Having other not curable cancers in the past 5 years, excluding the cured or treatable ones, such as basal skin carcinoma, squamous cell skin carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc;
6. Active autoimmune diseases required systemic treatment in the past 2 years, excluding vitiligo, type I diabetes, and autoimmune thyroiditis indued hypothyroidism that is curable by thyroid hormone replacement therapy;
7. Active tuberculosis (TB);
8. Confirmed infection of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
9. Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV):

   1. HBsAg positive and HBV DNA ≥ 1000 IU/mL;
   2. Positive test results of HCV RNA.
10. Women who are pregnant or breastfeeding;
11. Patients who are unavailable for venipuncture and/or intolerable for intravenous catheterization;
12. Interstitial lung disease;
13. History or basis of any clinically significant cardiovascular diseases as follows: abnormal electrocardiogram indicating additional risk for patients at the discretion of investigator; history of congestive heart failure (CHF) of grade III or above as documented by New York Heart Association (NYHA) criteria; history of cerebral infarction or myocardial infarction within 3 months prior to first dose; uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg); unstable angina; serious uncontrolled arrhythmia; baseline left ventricular ejection fraction (LVEF) < 50% or cardiac wall motion abnormalities identified by echocardiogram (ECHO).
14. Patients accepting other study drugs or anti-infective vaccine (e.g., influenza vaccine, and varicella vaccine) within 28 days prior to the first dose, and COVID-19 （Corona Virus Disease 2019）vaccine is permitted
15. Patients with anti-tumor vaccine therapy within 3 months prior to the first dose, and prophylactic HPV（human papilloma virus） vaccine is permitted;
16. Previous treatment with anti-CTLA-4 drugs;
17. Patients accepting systemic corticosteroids treatment at the doses of immunosuppressive effects (prednisone > 10 mg/day or equivalent level) within 2 weeks before the first dose; patients accepting immunosuppressive agents or glucocorticoids (at doses equivalent to prednisone > 10 mg/day) within 2 weeks before the first dose. Note: Epinephrine replacement therapy (equivalent to prednisone ≤ 10 mg/day) is allowed for patients without active immune disorder . Topical, intraocular, intra-articular, intranasal, and inhaled corticosteroids, which lead to (low systemic absorption, are allowed; short-term corticosteroids treatment is allowed for prophylactic therapy (e.g., be allergic to contrast media) or non-autoimmune diseases (e.g., delayed hypersensitivity reactions after exposure to allergens).
18. Patient accepting any antitumor traditional Chinese patent medicine within 2 weeks prior to the first dose (any antitumor traditional Chinese patent medicine is prohibited during this study).
19. Active infection requiring systematic treatment/antibiotics. Patient accepting intravenous anti-infective therapy with one week prior to the first dose or undergoing systematic anti-infective agents ≥ 7 days;
20. Received live attenuated vaccines within 4 weeks prior to the first dose, or plan to receive live attenuated vaccines during the study;
21. Allergic to any component of JS007;
22. Patients are not ineligible if meet at least one of the following conditions prior to the first dose :

    i. Major surgery requiring general anesthesia within 4 weeks prior to the first dose; ii. Surgery requiring local/epidural anesthesia within 72 hours prior to the first dose; iii. Skin biopsy requiring local anesthesia within 1 hour prior to the first dose.
23. Patients who are not appropriate for this trial due to other reasons at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to 12 approximately months
  The maximum tolerated dose (MTD) is defined as the highest dose at which DLT （Dose-Limiting Toxicity）occurs in <1/3 subjects
DLT | 21 days after first infusion of study drug
  DLT is defined as any of the specified toxicities evaluated as at least possibly related with the study drug within 21 days after the first dose (NCI-CTCAE v5.0)
Adverse Events | Up to 12 approximately months
  AE is assessed according to NCI-CTCAE 5.0
Serious Adverse Events | Up to 12 approximately months
  SAE（Serious adverse event） is assessed according to NCI-CTCAE 5.0
Incidence of immune-related adverse events (irAE) | Up to 12 approximately months
  IrAE is assessed according to NCI-CTCAE 5.0
severity of immune-related adverse events (irAE) | Up to 12 approximately months
  IrAE is assessed according to NCI-CTCAE 5.0

SECONDARY OUTCOMES:
peak concentration (Cmax) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters peak concentration (Cmax);
trough concentration (Ctrough) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters trough concentration (Ctrough)
time to peak (Tmax) | Up to 18 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters time to peak (Tmax);
area under the plasma drug concentration-time curve (AUC0-t ) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters area under the plasma drug concentration-time curve (AUC0-t )
area under the plasma drug concentration-time curve (AUC0-inf) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters area under the plasma drug concentration-time curve (AUC0-inf);
elimination half-life (t1/2) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters elimination half-life (t1/2)
clearance rate (CL) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters clearance rate (CL);
apparent volume of distribution(Vd) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; apparent volume of distribution(Vd)
volume of distribution (Vss) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters volume of distribution (Vss)
mean retention time (MRT) | Up to 12 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters mean retention time (MRT)
The number of lymphocyte in peripheral blood before and after administration | Up to 12 approximately months
  The number of lymphocyte in peripheral blood before and after administration
The proportion of lymphocyte in peripheral blood before and after administration | Up to 12 approximately months
  The proportion of lymphocyte in peripheral blood before and after administration
anti-drug body (ADA) | Up to 12 approximately months
  incidence of anti-drug body (ADA)
neutralizing antibody (Nab) | Up to 12 approximately months
  incidence of neutralizing antibody (Nab)
neutralizing antibody (Nab) | Up to 12 approximately months
  concentration of neutralizing antibody (Nab)

OTHER OUTCOMES:
ORR | Up to 12 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors), including objective response rate (ORR).
DOR | Up to 12 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors) , including duration of response (DOR);
DCR | Up to 12 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors) , including disease control rate (DCR);
PFS | Up to 12 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors) , including progression-free survival (PFS)
OS | Up to 12 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors) , including overall survival (OS);
CTLA-4（cytotoxic T lymphocyte-associated antigen-4） | Up to 12 approximately months
  Expression of CTLA-4 in tumor tissues before administration
FoxP3（transcription factor Forkhead box P3） | Up to 12 approximately months
  Expression of FoxP3 in tumor tissues before administration
IDO（(indoleamine 2,3-dioxy- genase） | Up to 12 approximately months
  Expression of IDO in tumor tissues before administration
mutation of immune related genes in tumor tissues before administration | Up to 12 approximately months
  mutation of immune related genes in tumor tissues before administration
expression of immune related genes in tumor tissues before administration | Up to 12 approximately months
  expression of immune related genes in tumor tissues before administration

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medical, Shanghai, China

REFERENCES:
- [Derived] Zhou C, Jiang J, Xiang X, Liu H, Wu G, Zeng R, Lu T, Zhang M, Shen Y, Hong M, Zhang J. Preclinical investigations and a first-in-human phase 1a trial of JS007, a novel anti-CTLA-4 antibody, in patients with advanced solid tumors. Exp Hematol Oncol. 2024 Oct 1;13(1):98. doi: 10.1186/s40164-024-00567-7. PMID 39354625